CLINICAL TRIAL: NCT04042337
Title: Improving Access to Pivotal Response Treatment (PRT) Via Telehealth Parent Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Grace Gengoux, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 52597
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRT Telehealth (Experimental): Participating parents will receive 12 weekly 60-minute parent training sessions via secure videoconference to learn Pivotal Response Treatment
  Interventions: Behavioral: Pivotal Response Treatment
- Waitlist (No Intervention): Participants will continue stable community-based treatments

INTERVENTIONS:
Behavioral: Pivotal Response Treatment — PRT will target functional communication abilities
  Arms: PRT Telehealth

SUMMARY:
There is an urgent need for improved access to effective autism treatments. With advances in technology, distance learning models have particular promise for families who cannot access evidence-based parent training locally or may be on long wait-lists for behavioral treatments. Pivotal Response Treatment (PRT) is an established treatment for autism spectrum disorder (ASD); however, a telehealth PRT model has not yet been evaluated in a controlled trial. This study will examine the effects of training parents in PRT via secure video conferencing and investigate 1) whether parents can learn via telehealth to deliver PRT in the home setting (PRT-T) and 2) whether their children will show greater improvement in functional communication skills compared to children in a waitlist control group. Participants will include 40 children age 2 to 5 years with ASD and significant language delay. Eligible children will be randomly assigned to either PRT-T (N=20) or waiting list (N=20). Weekly 60-minute parent training sessions will be delivered for 12 weeks via secure video conferencing software by a PRT-trained study therapist. The effects of PRT-T on parent fidelity of PRT implementation, child communication deficits including frequency of functional verbal utterances, and parent-report of communication skills on standardized questionnaires will be evaluated. This research will provide a foundation for wider dissemination of technology-based solutions to improve access to ASD treatment.

ELIGIBILITY:
Inclusion Criteria: Participants will include children ages a) 2:0 to 5:11 years, b) diagnosed with ASD (based on history, review of available medical records including diagnostic testing, e.g., ADOS) or suspicion of ASD diagnosis and confirmed with Autism Diagnostic Interview-Revised (ADI-R; completed by phone), c) with significant adaptive communication deficits (i.e., either a Vineland-3 Communication subscale 2SD below average for 2 and 3 year olds and 3 SD below for 4 and 5 year olds or a Vineland-3 Expressive V-scale Score 2 SD below average for 2 and 3 year olds, or 3 SD below for 4 and 5 year old, and at least moderate severity on the CGI-S language subscale), d) able to vocalize with communicative intent during home video observation, e) stable treatment for at least 2 weeks prior to baseline (e.g., ABA, special education) with no more than 60 minutes per week 1:1 speech therapy and no anticipated changes during study participation, and f) an English-speaking parent able to consistently participate in study procedures.

Exclusion Criteria.

a) children who have a primary language other than English, b) parent or child diagnosed with severe psychiatric disorder or unstable medical problem, c) child participating in >15 hours per week of 1:1 ABA treatment at home, d) unstable medical condition such as severe seizures, e) Severe behavioral difficulties (e.g., self-injury or aggression that could present a safety risk to the child or family members during implementation of the intervention), f) previous adequate trial of pivotal response treatment, or g) living within 200 miles of Stanford University.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2025-10-29 (Actual); Study Completion 2025-10-29 (Actual)

PRIMARY OUTCOMES:
Change in Parent Fidelity of PRT Implementation from Baseline to Week 12 | Baseline, Week 12
  Based on behavioral coding of parent-child interaction videos in the home

SECONDARY OUTCOMES:
Change in Child Frequency of Functional Utterances from Baseline to Week 12 | Baseline, Week 12
  Based on behavioral coding of parent-child interaction videos in the home

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry and Behavioral Sciences, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No